CLINICAL TRIAL: NCT03634683
Title: A Phase I/II, Open Label, Single Arm, Multicenter Study of LioCyx in Subjects With Recurrent Hepatitis B Virus-Related Hepatocellular Carcinoma Post Liver Transplantation
Brief Title: A Study of LioCyx in Patient With Recurrent HBV-related HCC Post Liver Transplantation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Major changes in manufacturing process and investigational product
Sponsor: Lion TCR Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-HCC-001
Record Dates: First submitted 2018-07-20; First posted 2018-08-16 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Recurrent Hepatocellular Carcinoma
Keywords: recurrent hepatocellular carcinoma; hepatitis B virus-related; post liver transplantation; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LioCyx (Experimental): This is a single-arm study.
  Patients will receive escalating doses of LioCyx on Day 1, Day 8, Day 15 and Day 22 of the first 28-day treatment cycle, followed by every 2-week dosing on Day 1, Day 15, Day 29 and Day 43 of repeated cycle. A 21-day treatment break will be given between each cycle.
  Interventions: Biological: LioCyx

INTERVENTIONS:
Biological: LioCyx — Autologous T cells transfected with mRNA encoding HBV antigen-specific TCR

SUMMARY:
Hepatocellular carcinoma (HCC) represent approximately 70-85% of liver cancer, in which Hepatitis B virus (HBV) is the major etiologic agent accounting for at least 80% of HCC in Asian countries. Overall, transplantation remains the best option however, HCC recurrence rate is high among liver transplant patients.

While there are limited treatment measures for HBV-related HCC recurrences, the study hypothesized that LioCyx is capable of lysing target liver cells expressing the HBV cognate antigens and provide clinical benefit to patients with HBV-related HCC.

DETAILED DESCRIPTION:
The study is a Phase I/II, open label, single-arm, multicenter study of LioCyx. Subjects with recurrent hepatitis B virus-related hepatocellular carcinoma who undergone liver transplantation will be enrolled.

Approximately 6-12 subjects will be enrolled in Phase 1 dose regimen exploration, and approximately 60 subjects will be enrolled to characterize the safety and evaluate the efficacy of LioCyx"

All subjects will be followed up for survival until death.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent locally advanced and/or metastatic hepatocellular carcinoma (HCC) post liver transplantation
* Life expectancy of 3 months or greater
* Have measurable disease by the revised response evaluation criteria in solid tumors (mRECIST)
* History of positive test for hepatitis B virus surface antigen (HBsAg)
* Expression of LioCyxTM target epitopes within specific human leukocyte antigen (HLA) class I profile
* Had received treatment with at least one standard therapy or refused, appropriate approved therapy for their disease
* 21 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Known, clinically suspected or has history of central nervous system (CNS) and bone metastasis
* Tumor burden in the liver exceeding 70%
* Significant ongoing immunologic rejection based on pathology and clinical diagnosis
* Evidence or history of significant bleeding diathesis or coagulopathy
* Prior exposure to any cell therapy such as, but not limited to NK, CIK, DC, CTL, stem cells therapy
* Known history of testing positive for human immunodeficiency virus (HIV) 1 or 2 or known acquired immunodeficiency syndrome (AIDS)
* Lack of peripheral venous or central venous access or any condition that would interfere with drug administration or collection of study samples
* Women who are pregnant or breast-feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Safety based on Incidence of Treatment-Emergent Adverse Events (AEs) and Serious AEs | Start of Treatment until 28 days post last dose
  Review the safety profile of LioCyx by assessing the incidence of AEs and SAEs

SECONDARY OUTCOMES:
Overall Response Rate | Start of Treatment until first documented CR or PR, assessed up to 62 treatment weeks (protocol-defined treatment duration is until disease progression, death, or loss to follow up, whichever came first)
  Tumor assessment will be according to mRECIST. This is based on percentage of participants with Complete Response (CR) and Partial Response (PR) according to mRECIST from baseline.
Overall Survival according to mRECIST | Start of Treatment until first protocol-defined PD, and survival follow up until death, assessed up to 62 treatment weeks (protocol-defined treatment duration is until disease progression, death, or loss to follow up, whichever came first)
  Assess the efficacy following LioCyx in prolonging overall survival of patients in HBV-related HCC patients
Quality of life of patients | Baseline to 28 days post treatment (end of treatment)
  Compare the quality of life of patients based on [Functional Assessment of Chronic Illness Therapy- Hepatobiliary (FACIT-Hep), version 4]

CONTACTS AND LOCATIONS:
Locations (3):
- China (2):
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangzhou
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangzhou
- National University Hospital, Singapore, Singapore